CLINICAL TRIAL: NCT05747677
Title: A Single-Arm Clinical Study Evaluating the Efficacy of Post-Exposure Prophylaxis , Safety, and Tolerability of HH-120 Nasal Spray in Close Contacts of SARS-CoV-2
Brief Title: A Study of HH-120 Nasal Spray in Close Contacts of Those Diagnosed With COVID-19
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Beijing Ditan Hospital (Other)
Responsible Party: Principal Investigator, Ronghua Jin, Chief Physician, Beijing Ditan Hospital
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Prevention
Other Study IDs: HH120-IIT-NS01
Record Dates: First submitted 2023-02-24; First posted 2023-02-28 (Actual); Last update posted 2023-02-28 (Actual); Status verified 2023-02

CONDITIONS: COVID-19; SARS-CoV-2 Infection
MeSH Terms: conditions — COVID-19

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- HH-120 Nasal Spray (Experimental)
  Interventions: Drug: HH-120 Nasal Spray

INTERVENTIONS:
Drug: HH-120 Nasal Spray — HH-120 nasal spray, 1 spray to each nostril of the participant each time,8-10 times per day, until the discharge of the SARS-CoV-2 infected patients or confirmed infection of the participant, whichever occurs first.

SUMMARY:
This study is to evaluate the efficacy of post-exposure prevention and safety of HH-120 nasal spray in participants who are caregivers of hospitalized patients infected with SARS-CoV-2. HH-120 nasal spray are administrated 8-10 times to the participants per day until the discharge of the SARS-CoV-2 infected patients or confirmed infection of the participant, whichever occurs first.

ELIGIBILITY:
Inclusion Criteria:

* Male and female subjects aged 18 or above;
* Caregivers of hospitalized children who are infected with SARS-CoV-2;
* Negative qRT-PCR nucleic acid test result during the screening;
* Willing and able to give written informed consent.

Exclusion Criteria:

* Those who have child-bearing plan or are unable to voluntarily take effective contraceptive measures, or plan to donate sperm/ovum during the study or within 3 months after the end of the study;
* Female subjects who are positive for human chorionic gonadotropin (β-Human Chorionic Gonadotropin, β-HCG) or are breastfeeding;
* Have used antiviral drugs with a therapeutic effect on COVID-19 within 3 months before screening, including various monoclonal antibodies (tixagevimab and cilgavimab, tocilizumab, ambavirumab and romisvir, Bamlanivimab, Etesevimab, Bebtelovimab, Casirivimab and imdevimab, Sotrovimab), convalescent plasma, hydroxychloroquine, Paxlovid (Nimatevir/ritonavir), Azvudine, Baricitinib, molnupiravir, remdesivir, interference drug, ribavirin, arbidol and lopinavir, etc.; (except those with the wash-out time longer than 5 half-lives);
* Those who have participated in clinical trials of SARS-CoV-2 neutralizing antibodies or participated in clinical trials of other drugs within 4 weeks before screening;
* Those who have a history of severe allergies or are sensitive to inhaled allergens; or are known to be sensitive to the ingredients of the study drug, other monoclonal antibody drugs, and therapeutic protein preparations (fresh or frozen plasma, human serum albumin, cytokines, interleukin, etc.) Factors, etc.) have allergies or hypersensitivity reactions;
* Those who have received the COVID-19 vaccine within 2 weeks before the study drug administration or plan to receive the COVID-19 vaccine during the study;
* Those who cannot tolerate with nasal spray treatment;
* Any other circumstances that the researchers deemed not suitable for participating in the study.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 14 (Actual)
Dates: Start 2022-06-14 (Actual); Primary Completion 2023-02-06 (Actual); Study Completion 2023-02-06 (Actual)

PRIMARY OUTCOMES:
The proportion of subjects infected with SARS-CoV-2 | As of the discharge of the SARS-CoV-2 infected patients, an average 1 week

SECONDARY OUTCOMES:
The incidence and severity of adverse events and the serious adverse events | As of the 7th day after the last study drug administration

CONTACTS AND LOCATIONS:
Locations (1):
- Beijing Ditan Hospital,Capital Medical University, Beijing, Beijing Municipality, China